CLINICAL TRIAL: NCT06034873
Title: Comparative Study Between Ultrasound Guided Pericapsular Nerve Block Versus iv Sedation Analgesia in Reduction of Shoulder Dislocation, Double Blinded Controlled Randomized Clinical Trial
Brief Title: Ultrasound Guided Pericapsular Nerve Block Versus iv Sedation Analgesia in Reduction of Shoulder Dislocation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Abdel Fatah, lecturer of anaesthesia, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC 17-7-2023
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2023-10

CONDITIONS: Perioperative Pain
MeSH Terms: interventions — Propofol; Fentanyl; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): In the IVAS group, the patients intravenous propofol combined with fentanyl. The sequence will be to inject fentanyl 1 μg•kg-1•min-1 first within 1 min and then inject propofol 2 mg•kg-1•min-1.
  Interventions: Drug: Propofol injection and fentanyl
- Group B (Active Comparator): Patients will be anesthetized with ultrasound-guided pericapsular nerve group block (PENG block) using 20 ml of 0.25% bupivacaine.
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Propofol injection and fentanyl — The sequence will be to inject fentanyl 1 μg•kg-1•min-1 first within 1 min and then inject propofol 2 mg•kg-1•min-1.
  Other Names: deprivan
  Arms: Group A
Drug: Bupivacain — Patients will be anesthetized with ultrasound-guided pericapsular nerve group block (PENG block) using 20 ml of 0.25% bupivacaine.
  Other Names: markain
  Arms: Group B

SUMMARY:
When someone experiences a shoulder dislocation, it can be extremely painful. Emergency physicians often choose to use conscious sedation to help reduce the pain. However, some patients may not be able to tolerate conscious sedation due to concerns about their ability to breathe properly or the risk of inhaling fluids. A recently developed technique called Ultrasound-guided Pericapsular Nerve Group (PENG) block is used to block the articular branches of the shoulder and the pericapsular spread around the glenohumeral joint. The PENG block is commonly used in hip surgery and is effective in providing motor-sparing analgesic results.

DETAILED DESCRIPTION:
When someone experiences a shoulder dislocation, it can be extremely painful. Emergency physicians often choose to use conscious sedation to help reduce the pain. However, some patients may not be able to tolerate conscious sedation due to concerns about their ability to breathe properly or the risk of inhaling fluids. In an ideal scenario, the surgeon could achieve complete pain control and muscle relaxation without compromising the patient's airway. There are various techniques available to facilitate shoulder reduction, including interscalene block, general anesthesia, and intravenous analgesia. All of these methods can help the surgeon ease the patient's pain and reduce the likelihood of complications.1 When choosing the anesthesia method for reducing ASD, the top priority is ensuring the patient's comfort through pain management. The anesthesia helps to relax the muscle spasms, making it easier to reduce the ASD. The goal is to relocate the shoulder with minimal risk of complications.

A recently developed technique called Ultrasound-guided Pericapsular Nerve Group (PENG) block is used to block the articular branches of the shoulder and the pericapsular spread around the glenohumeral joint. The PENG block is commonly used in hip surgery and is effective in providing motor-sparing analgesic results.

ELIGIBILITY:
Inclusion Criteria:

* (ASA )classes I and II
* patients of either sex, above the age of 18
* patients will undergo dislocated shoulder

Exclusion Criteria:

* the patient's refusal to participate
* coagulation disorders
* allergy to local anesthetic
* history of daily opioid intake
* patients with cognitive impairments

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
length of hospital stay | 1st 24 hours
  the period when the patient stayed in the hospital

SECONDARY OUTCOMES:
reduction time | 1st hour after intervetion
  the period from the beginning to the end of reduction
the visual analogue scale(VAS) | 30 minutes ,2,4,8,12 hours postoperative
  ranges from 0 to 10, with 0 representing no pain and 10 being the most intense pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ah Abdelfatah, MD, Principal Investigator — banha faculity of medicine
Locations (1):
- Banha faculity of medicine, Banhā, Elqalyoubea, Egypt